CLINICAL TRIAL: NCT01915433
Title: Wahls Paleo Diet and Progressive Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terry L. Wahls (Other)
Responsible Party: Sponsor-Investigator, Terry L. Wahls, Study Director, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201302829
Record Dates: First submitted 2013-07-25; First posted 2013-08-02 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Multiple Sclerosis
Keywords: Secondary Progressive Multiple Sclerosis; Primary Progressive Multiple Sclerosis; Relapsing progressive multiple sclerosis; relapsing remitting multiple sclerosis; Fatigue; Quality of life; Paleo; Nutrition; Ketogenic
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis, Relapsing-Remitting; Fatigue | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Wahls Paleo Plus (Experimental): Wahls Paleo Plus diet (ketogenic diet)
  Interventions: Other: Wahls Paleo Plus
- Wahls Diet (Experimental): Wahls Diet (modified paleolithic diet)
  Interventions: Other: Wahls Diet
- Usual Care (No Intervention): Control - usual care only.

INTERVENTIONS:
Other: Wahls Paleo Plus — The study diet is based upon a Paleolithic Diet, also known as a Hunter Gatherer Diet, which exceeds the recommended daily allowance of water soluble vitamins and minerals 1.5 to 8 fold and improves lipids, inflammatory biomarkers and blood pressure. The study diet is further structured to be a low in carbohydrate and high in fat but still ensure consumption of the specific micronutrients important to optimal brain function. This diet is designed to induce a low level nutritional ketosis.
  Other Names: Wahls Paleo Plus (ketogenic diet)
  Arms: Wahls Paleo Plus
Other: Wahls Diet — The study diet is based upon a Paleolithic Diet, also known as a Hunter Gatherer Diet, which exceeds the recommended daily allowance of water soluble vitamins and minerals 1.5 to 8 fold and improves lipids, inflammatory biomarkers and blood pressure. The study diet is further structured to be a low glycemic diet and also ensure consumption of the specific micronutrients important to optimal brain function.
  Other Names: Wahls Diet (modified paleolithic diet)
  Arms: Wahls Diet

SUMMARY:
Based on favorable preliminary data from ongoing studies testing the safety and tolerability of a nutrition, exercise and neuromuscular electrical stimulation funded by Direct MS, the investigators are proposing a pilot study focused on the Wahls Paleo plus Diet and Wahls Diet intervention to usual care. The intent is to measure the effect size of a Wahls Paleo plus Diet and the effect size of the Wahls Diet in reducing fatigue and improving quality of life scores as measured by fatigue severity scale score and MS quality of life 54 physical and mental scores and various subscale scores. Inclusion criteria is the presence of fatigue and the diagnosis secondary and primary progressive MS, progressive relapsing MS or relapsing-remitting MS with an expanded disability status scale score (EDSS) score of 4.5 or greater but otherwise stable medically. The Wahls Paleo plus (ketogenic diet) and the Wahls diet (modified paleolithic diet) groups will be instructed in completing a daily food log and receive coaching from registered dieticians who are expert in motivational interviewing. The control group will receive usual care. Biomarkers of nutrient levels (e.g. vitamin) and inflammation, blood sugar and insulin levels will be monitored. Additional blood will be frozen for future analysis. Nutrient (e.g. vitamin and antioxidant) intake will be assessed using food frequency questionnaires and 24 hr diet recalls. Test of endothelial function will be done at baseline and 12 weeks. Outcome measures will be change in quality of life and fatigue, endothelial function and blood biomarkers between enrollment and end of study at 12 weeks. The hypotheses are that the diet intervention groups will experience reduced fatigue and improved quality of life and improved biomarkers 1) between zero and 12 weeks and that the wahls paleo plus (ketogenic diet) and the wahls diet (modified paleolithic diet) groups will experience more improvements in quality of life and reduced fatigue and in biomarkers than the usual care group experiences at 12 weeks. The usual care group will be given instruction in following both the wahls paleo plus and the wahls diet plans and how to utilize the daily food logs at the end of study visit. The usual care group will receive one nutrition coaching call to assist with implementation of the study diet.

DETAILED DESCRIPTION:
Specific Aim 1. To assess changes in fatigue severity (primary outcome measure) and quality of life, motor, cognitive and emotional functions (secondary measures) the intervention groups (wahls paleo plus and wahls diet group)to usual care.

Hypothesis 1a: The Wahls Paleo plus group and the wahls diet group will both demonstrate more improvements in quality of life and fatigue between baseline and 12 weeks than usual care group.

Hypothesis 1b. The wahls paleo plus group will demonstrate more improvement in quality of life and fatigue than the wahls diet group.

Specific Aim 2. To assess changes in the blood biomarkers and endothelial function as the subject progresses through the study interventions.

Hypothesis 2a: The wahls paleo plus and the wahls diet group will demonstrate more favorable changes in blood biomarkers obtained at baseline and week 12 than the usual care group.

Hypothesis 2b: The wahls paleo plus group will demonstrate more favorable changes in blood biomarkers and quality of life than the wahls diet group experiences obtained at baseline and week 12.

Hypothesis 2c: The wahls paleo plus and the wahls diet group will demonstrate more favorable changes in measures of endothelial function between baseline and week 12 than will be observed in the usual care group.

Hypothesis 2d: The wahls paleo plus will demonstrate more favorable changes in measures of endothelial function between baseline and week 12 than the wahls diet group.

ELIGIBILITY:
Inclusion Criteria - to complete 2 week RUN IN to determine eligibility for Main Study:

Inclusion Criteria -

1. Secondary or Primary Progressive MS, relapsing progressive MS, relapsing- remitting MS
2. Generally able to walk 25 feet in less than 60 seconds;
3. significant fatigue as documented by a fatigue severity scale score of 4 or more OR a modified fatigue impact scale score of 38 or higher.
4. age between 30 and including 65 at entry into the RUN IN study,
5. non smoker,
6. willingness to be randomized
7. Mild gait disability as shown by an EDSS score of 4.5 or higher
8. Confirmed MS diagnosis using McDonald criteria
9. Eating standard American diet.

Exclusion Criteria for RUN IN to determine eligibility:

1. change in medication in the prior 90 days, taking anti-platelet or anticoagulant therapy therapy, or having a major psychiatric disorder making compliance difficult,
2. SELF REPORTED history of current diagnosis of diabetes, or active liver, kidney or clinically significant heart disease,
3. unable to record daily weight at home,
4. eating a vegetarian diet or chronic diarrhea, have already adopted a Paleo Diet (as defined by a complete elimination of grain, dairy, and legumes)
5. unable to cope with 30% in grocery bill,
6. Alanine aminotransferase value > 2X normal, or elevated creatinine value, (main study only)
7. incompetence.
8. Too low or too high BMI.
9. Inability to follow study diet, which requires shopping carefully and food preparation, by either the study subject or with the help of an adult companion to do the shopping and food preparation.
10. aversion to coconut milk

Main Study Inclusion Criteria

1) Successful completion of RUN IN Study - which means, the subject completed the various quest. and survey documents that are part of the RUN-IN study, completed the food diary for each day they participated in the RUN-IN, the subject is eating the standard American Diet as documented by the daily food logs and the 24 hour dietary recalls.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Perceived Fatigue | Baseline, weeks, 4,8 and 12
  Fatigue as measured by the fatigue severity scale and the modified fatigue impact scale

SECONDARY OUTCOMES:
Biomarkers | Baseline and 12 weeks
  Biomarkers include weight, Body Mass Index,and blood biomarkers of renal and liver function, vitamin levels (A,C,K,D, B vitamins), homocysteine, h.s. c- reactive protein (CRP)
Biomarkers - glucose and ketones | Baseline and at 4, 8, 12 weeks
  GLucose, insulin, ketones, hemoglobin a1c to assess insulin sensitivity. Full intervention at baseline, and weeks 4,8,12 Minimal intervention at baseline and week 12.
24 hr food recalls. | Baseline and 12 weeks
  The 24 hr recalls will be collected at baseline in in the last 4 weeks of study. This will include nutrient analyses as well.
Daily Food logs | Baseline through end of study (12 weeks)
  This is a record of daily food and beverage consumption. The two intervention groups will keep the record daily. The usual care group will keep the a food record the initial two weeks and for two weeks between weeks 10 and 12.
MS functional composite score. | Baseline and end of study (12 weeks)
  This a composite of tests involving tests of walking, hand coordination and mental addition.
6 minute walk test | Baseline and week 12
  Subject will walk 6 minutes. They may rest as needed during the 6 minute time period. The total length of time that is walked will be recorded.
Medical symptoms quest. (MSQ) | Baseline, weekly through week 12
  Scored review of systems questionaire
Life spaces score | Baseline and week 12
  Questions about the locations subjects has been in the prior time period of interest.
Medication audit | Baseline
  List of currently used medications, vitamins, supplements and over the counter medications.
Physical examination | baseline and 12 weeks
  Summary of physical findings from physical examination.
Health questions | baseline
  A list of questions to identify common medical comorbid conditions and their severity if present.
MS Quality of Life (MSQoli 54) | Baseline, week 12
  MS Qoli 54 is a series of questions about physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life.
MS Quality of life inventory (MSQLI) | Baseline and week 12
  MSQLI is a series of questions asking about daily life. Includes physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life.
Demographic data | Baseline and week 12
  Questions about demographic attributes such as race, education, handedness.
Functional Medicine assessment summary | Baseline or 12 weeks
  A series of questions about a number of environmental risk factors for development of neurological and medical symptoms. Completed prior to orientation to study intervention diet after randomization (intervention groups) or at 12 weeks for usual care group.
Veteran Specific Activity Quest. | Baseline and 12 weeks.
  Series of questions about the tasks of daily life to identify how much activity the individual can safely do.
MS Function Scale | baseline and week 12
  A series of questions about the tasks of daily life.
Satiety scale | Baseline and weeks 10 and 11
  A series of questions about the sense of satiety or sense of fullness.
Harvard Food Frequency Quest. | Baseline
  A series of questions about the frequency of a variety of foodstuffs to estimate nutrient intake.
Brachial artery dilation (FMD)and endothelium-dependent dilation, EDD) and endothelium-independent dilation | Baseline and week 12
  Brachial artery FMD and endothelium-independent dilation will be determined non-invasively using high-resolution ultrasonography.
Expanded disability status score | Baseline and 12 weeks
  Assessment of disability status

CONTACTS AND LOCATIONS:
Overall Officials: Terry L Wahls, MD, Study Director — University of Iowa
Locations (1):
- Univeristy of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wahls TL, Reese D, Kaplan D, Darling WG. Rehabilitation with neuromuscular electrical stimulation leads to functional gains in ambulation in patients with secondary progressive and primary progressive multiple sclerosis: a case series report. J Altern Complement Med. 2010 Dec;16(12):1343-9. doi: 10.1089/acm.2010.0080. PMID 21138391
- [Background] Reese D, Shivapour ET, Wahls TL, Dudley-Javoroski SD, Shields R. Neuromuscular electrical stimulation and dietary interventions to reduce oxidative stress in a secondary progressive multiple sclerosis patient leads to marked gains in function: a case report. Cases J. 2009 Aug 10;2:7601. doi: 10.4076/1757-1626-2-7601. PMID 19918474
- [Background] Wahls TL. The seventy percent solution. J Gen Intern Med. 2011 Oct;26(10):1215-6. doi: 10.1007/s11606-010-1631-3. No abstract available. PMID 21253878
- [Background] Riccio P. The molecular basis of nutritional intervention in multiple sclerosis: a narrative review. Complement Ther Med. 2011 Aug;19(4):228-37. doi: 10.1016/j.ctim.2011.06.006. Epub 2011 Jul 27. PMID 21827937
- [Background] Bourre JM. Effects of nutrients (in food) on the structure and function of the nervous system: update on dietary requirements for brain. Part 2 : macronutrients. J Nutr Health Aging. 2006 Sep-Oct;10(5):386-99. PMID 17066210
- [Background] Bourre JM. Effects of nutrients (in food) on the structure and function of the nervous system: update on dietary requirements for brain. Part 1: micronutrients. J Nutr Health Aging. 2006 Sep-Oct;10(5):377-85. PMID 17066209
- [Background] Bowman GL, Silbert LC, Howieson D, Dodge HH, Traber MG, Frei B, Kaye JA, Shannon J, Quinn JF. Nutrient biomarker patterns, cognitive function, and MRI measures of brain aging. Neurology. 2012 Jan 24;78(4):241-9. doi: 10.1212/WNL.0b013e3182436598. Epub 2011 Dec 28. PMID 22205763
- [Background] Frassetto LA, Schloetter M, Mietus-Synder M, Morris RC Jr, Sebastian A. Metabolic and physiologic improvements from consuming a paleolithic, hunter-gatherer type diet. Eur J Clin Nutr. 2009 Aug;63(8):947-55. doi: 10.1038/ejcn.2009.4. Epub 2009 Feb 11. PMID 19209185
- [Background] Stafstrom CE, Rho JM. The ketogenic diet as a treatment paradigm for diverse neurological disorders. Front Pharmacol. 2012 Apr 9;3:59. doi: 10.3389/fphar.2012.00059. eCollection 2012. PMID 22509165